CLINICAL TRIAL: NCT04663399
Title: IMMunological resPonse Assessment afteR Acute iSchemic Stroke Treated With Endovascular Therapy
Brief Title: IMMunological resPonse Assessment afteR Acute iSchemic Stroke Treated With Endovascular Therapy (IMPRESS)
Acronym: IMPRESS
Status: Recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: BMR_2020_32
Record Dates: First submitted 2020-11-25; First posted 2020-12-11 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Ischemic Stroke; Thrombectomy
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Each blood sample consists of 3x3 mL Citrate + 1x4 mL EDTA + 1x4 mL Heparin + 1x5 mL dry tube.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient with MT: Patients indicated for mechanical thrombectomy and benefiting from the procedure
  Interventions: Other: Prospective patient
- Patient without MT: Patients indicated for mechanical thrombectomy but not benefiting from the intervention due to clinical improvement (patients responding to thrombolysis)
  Interventions: Other: Prospective patient

INTERVENTIONS:
Other: Prospective patient — The immuno-inflammatory and thrombo-inflammatory profiles will be evaluated at inclusion, and at 24 hours +/- 12 hours of the reperfusion treatment.

SUMMARY:
IMPRESS study aims to describe the immuno-inflammatory and thrombo-inflammatory profiles during the first 24/36 hours of treatment of patients suffering from AIC treated with TM, and to study the possible impact of these profiles on the functional prognosis at 3 and 12 months of AIC treatment.

DETAILED DESCRIPTION:
Stroke is the second leading cause of death worldwide, the leading cause of acquired disability and the second leading cause of dementia. Ischaemic strokes account for 80% of strokes, 40% of which are caused by occlusion of a large-calibre artery in the polygon of Willis. In 2020, the treatment focuses on recanalisation, as quickly as possible. This is achieved medically by intravenous thrombolysis (IVT) and, since 2015, by mechanical thrombectomy (MT) in cases of proximal anterior artery occlusion. Thrombectomy has revolutionised the management of AIC, as it results in over 90% recanalisation at the end of treatment. However, more than half of patients managed between 3 and 6 hours, and recanalised with TM, remain dependent at 3 months.

In recent years, numerous studies (mainly preclinical) have highlighted the impact of the systemic and cerebral inflammatory reaction following AIC. Interestingly, this immuno-inflammatory reaction seems to follow a precise chronology and involves various immune players. Several preclinical studies in rodents have shown that this immunoinflammatory response appears to be strongly associated with prognosis (final stroke volume, disability and post-stroke dementia).

The absence of reliable biomarkers in humans to better describe and assess the chronology of the immuno-inflammatory profile after stroke appears to be a fundamental limitation to the introduction of innovative treatments. These biomarkers would make it possible to select and accurately assess the time required to introduce treatments such as immunomodulatory therapies (Natalizumab, Fingolimod, Copaxone, cell therapy, etc.). New studies seem necessary to identify peripheral biomarkers of the immuno-inflammatory state (cytokines, precise cell typing), and of thrombo-inflammation (NETose markers, neutrophil markers) and their consequences on disability after an ACI.

The aim of the IMPRESS study is therefore to describe the immuno-inflammatory and thrombo-inflammatory profiles during the first 24 +/-12 hours of the management of patients suffering from AIC treated with TM, and to study the possible impact of these profiles on the functional prognosis 3 and 12 months after the AIC has been managed.

ELIGIBILITY:
Inclusion Criteria:

* Patient with an acute ischemic stroke for which treatment with mechanical thrombectomy is indicated, whether or not thrombectomy is performed,
* Having received informed information about the study and having signed a consent to participate in the study (if this is not possible: information and consent of the trusted support person or family member if present; emergency inclusion if absent);
* Affiliated or beneficiary of a social security scheme or equivalent.

Non inclusion Criteria:

* Pregnant or breast-feeding women
* Patient benefiting from a legal protection measure

Exclusion Criteria:

None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for a mechanical thrombectomy as part of an acute ischemic stroke will be able to participate in the study.
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2023-02-23 (Actual); Primary Completion 2028-05-23 (Estimated); Study Completion 2028-05-23 (Estimated)

PRIMARY OUTCOMES:
Immuno-inflammatory and thrombo-inflammatory profiles in patients suffering from AIC and treated with mechanical Thrombectomie. | 21 months
  Blood plasma collected from patients at inclusion, and at 24 hours +/- 12 hours of the reperfusion treatment will be used to discover and validate panels of inflammatory biomarkers that are predictive of therapeutic response. The biomarkers will be measured using a multiplex preconfigured panels for inflammatory biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Maier, MD, Principal Investigator — Fondation Ophtalmologique Adolphe de Rothschild
Locations (1):
- Hôpital Fondation Adolphe de Rothschild, Paris, Paris, France